CLINICAL TRIAL: NCT02954237
Title: AMPLATZER™ Cardiac Plug Observational Post-Approval Study
Acronym: ACP China
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: SJM-CIP-CRD 881; SJM-CIP-10153 (Other: Abbott Medical (Note:protocol ID shown in Abbott system))
Record Dates: First submitted 2016-10-10; First posted 2016-11-03 (Estimated); Results first posted 2022-06-24 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Non-valvular Atrial Fibrillation (NVAF)
Keywords: Non-valvular atrial fibrillation (NVAF); Anticoagulant; Warfarin; Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- AMPLATZER™ Cardiac Plug: Subjects who were implanted with AMPLATZER™ Cardiac Plug will be included in this arm.
  Interventions: Device: AMPLATZER™ Cardiac Plug

INTERVENTIONS:
Device: AMPLATZER™ Cardiac Plug — The AMPLATZER™ Cardiac Plug is a transcatheter, self-expanding device intended for use in preventing thrombus embolization from the left atrial appendage. The device is constructed from a nitinol mesh and consists of a lobe and a disc connected by a central waist. The device is designed to facilitate occlusion. The lobe has stabilizing wires to improve device placement and retention. The device has threaded screw attachments at each end for connection to the delivery and loading cables. The device has radiopaque markers at each end and at the stabilizing wires. Device Sizes: 16, 18, 20, 22, 24, 26, 28, and 30 mm (lobe diameter) Delivery System: AMPLATZER TorqVue® 45º x 45º (sheath sizes 9, 10, or 13 Fr)

SUMMARY:
The purpose of this study is to observe the safety and effectiveness of the AMPLATZER™ Cardiac Plug (ACP) device in Chinese population indicated for use of AMPLATZER™ Cardiac Plug after its market approval by China FDA (CFDA). This is a prospective, multi-centre, single arm, post approval, observational study. The clinical study will be conducted at up to 35 sites in China. Approximately 343 subjects will be enrolled in this study.

The total study duration is expected to be approximately 7 years. The study population included patients who have non-valvular atrial fibrillation (NVAF) and are contraindicated to long-term oral anticoagulant; or patients who experience stroke or other thromboembolic event despite taking warfarin.

Scheduled office visits occur at 45 days (+45 days), 6M (+/- 3 weeks) 12M (+/- 6 weeks) and 24 M(+/- 6 weeks) post procedure; Phone contact follow up visits occur at, 36 M (+/- 6 weeks), 48M (+/- 6 weeks) and 60 M (+/- 6 weeks) post procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Patient who meets the current indications and per physician discretion for ACP implant
2. Patient who is ≥ 18 years of age at the time of enrolment
3. Patient who is able to provide written Informed Consent prior to any study related procedures

Exclusion Criteria:

1. Patient who is unable to comply with the follow-up schedule
2. Patient with the presence of intracardiac thrombus
3. Patient with active endocarditis or other infections producing bacteraemia
4. Patient who has low risk of stroke (CHA2DS2-VASC score is 0 or 1) or low risk of bleeding (HAS-BLED score<3)
5. Patient where placement of the device would interfere with any intracardiac or intravascular structures
6. Patient who is under medical conditions not appropriate to participate in the study in the opinion of the investigator
7. Patient with LAA anatomy that does not accommodate a device per the sizing guidelines
8. Patient who has a life expectancy of less than 2 years due to any condition
9. Patient who are currently participating in a clinical investigation that includes an active treatment arm
10. Patient who already had a left atrial appendage closure device implanted prior to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have non-valvular atrial fibrillation (NVAF) and are contraindicated to long-term oral anticoagulant; or patients who experience stroke or relevant event despite taking warfarin.
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2016-11-14 (Actual); Primary Completion 2021-01-29 (Actual); Study Completion 2021-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maren Wagner, Study Director — Abbott
Locations (6):
- China (6):
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Sir Run Run Shaw Hospital, Zhejiang, Hangzhou
  - Wuhan Asia Heart Hospital, Wuhan, Hubei
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Ningbo First Hospital, Ningbo, Liuting Saint
  - The First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 94 subjects were consented, and 91 were enrolled in the study. The first and last Amplatzer Cardiac Plug implants as part of the study occured on 14-Nov-2016 and 12-Mar-2019, respectively. The final 24-month follow-up visit occurred on 29-Jan-2021.
Period: Overall Study
Arm/Group | AMPLATZER™ Cardiac Plug
Started | 91
Completed | 48
Not Completed | 43
Not completed — Withdrawal by Subject | 25
Not completed — Missed visit | 16
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | AMPLATZER™ Cardiac Plug
Number analyzed (Participants) | 91
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.6 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 56
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  China | 91
HAS-BLED Score [Mean (Standard Deviation); unit: scores on a scale] — HAS-BLED scale is a scoring system that includes a set of questions to assess the level of risk for bleeding events. The total score ranges from 0 to 9 where a score of 0 indicates low risk, 1-2 indicates moderate risk, and ≥3 indicates high risk.
  scores on a scale | 3.5 (0.7)

OUTCOME MEASURES:

1. Primary Outcome: Short-Term Safety Endpoint: Composite Rate of Death, Stroke, Systemic Embolism, and Procedure or Device-related Complications Requiring Intervention
Description: The primary short-term safety endpoint was the composite of death, stroke (ischemic or haemorrhagic), systemic embolism and procedure or device-related complications requiring major cardiovascular or endovascular intervention.
Time Frame: Within 7 days of the procedure
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AMPLATZER™ Cardiac Plug
Number analyzed (Participants) | 91
percentage of participants | 1.1 [0.03 to 5.97]

2. Primary Outcome: Long-Term Safety Endpoint: Composite Rate of Device Embolization/Device Erosion/Device Interference With Surrounding Structure/Device Thrombus/Device Fracture/Device Infection/Device Perforation/Device Laceration/Device Allergy
Description: The primary long-term safety endpoint was the composite of of device embolization, device erosion, clinically significant device interference with surrounding structure, device thrombus, device fracture, device infection (endocarditis and pericarditis), device perforation, device laceration, or device allergy.
Time Frame: Within 2 years of the procedure
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AMPLATZER™ Cardiac Plug
Number analyzed (Participants) | 91
percentage of participants | 2.2 [0.57 to 8.69]

3. Primary Outcome: Long-Term Effectiveness Endpoint: Composite Rate of Ischemic Stroke or Systemic Embolism
Description: The primary long-term effectiveness endpoint was the composite rate of ischemic stroke or systemic embolism.
Time Frame: Within 2 years of the procedure
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AMPLATZER™ Cardiac Plug
Number analyzed (Participants) | 91
percentage of participants | 1.1 [0.16 to 7.54]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | AMPLATZER™ Cardiac Plug
All-Cause Mortality (participants affected / at risk) | 3/91
Serious Adverse Events (participants affected / at risk) | 28/91
Other Adverse Events (participants affected / at risk) | 0/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AMPLATZER™ Cardiac Plug (N=91)
Angina pectoris (Cardiac disorders) | 2
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cholelithiasis (Gastrointestinal disorders) | 1
Chronic Obstructive Pulmonary Disease (COPD) (Respiratory, thoracic and mediastinal disorders) | 2
Congestive Heart Failure (Cardiac disorders) | 3
Facial Paresis (General disorders) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Gastrointestinal Bleeding (Gastrointestinal disorders) | 1
Heart Failure (Cardiac disorders) | 3
Hemangioma (Blood and lymphatic system disorders) | 1
Intracerebral Haemorrhage (Blood and lymphatic system disorders) | 1
Pericardial Effusion (Cardiac disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3
Post-Menopausal Bleeding (Reproductive system and breast disorders) | 1
Seizure/Convulsions/Epilepsy (Nervous system disorders) | 1
Sinus Bradycardia/Sinus Bradycardia (Cardiac Arrhythmia) (Cardiac disorders) | 2
Stroke (Nervous system disorders) | 1
Subdural Haemorrhage (Vascular disorders) | 1
Thrombus on Device (Injury, poisoning and procedural complications) | 1
Unmasking Old Stroke Symptoms (Nervous system disorders) | 1
VASC Hematoma (Blood and lymphatic system disorders) | 1
Vertigo (Nervous system disorders) | 1
Other - Anaphylactic Shock (General disorders) | 1
Other - Arrhythmia (Cardiac disorders) | 1
Other - Pancytopenia (Blood and lymphatic system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-04): https://cdn.clinicaltrials.gov/large-docs/37/NCT02954237/Prot_SAP_000.pdf